CLINICAL TRIAL: NCT02099838
Title: The Randomized Multiple Center Trial for The Effectiveness and Safety of Adding Compound Preparation of Pioglitazone and Metformin for Type 2 Diabetic Patients Who Have Bad Glycemic Control With the Initial Treatment of Sulfonylureas
Brief Title: Effectiveness and Safety of Adding Compound Preparation of Pioglitazone and Metformin for Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Iron and Steel Workers' Hospital (Other); Wuhan Pu-Ai Hospital (Other); Hubei Xinhua Hospital (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Director of Department of Endocrinology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Tongji201202
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pioglitazone; Metformin; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone and Metformin (Experimental): Type 2 diabetic patients only took SUs previously. During a week for washout before the trial, they received diet and sport instructions, kept the SUs unchanged and didn't use any drugs affecting blood glucose. All participants added 1 tablet of pioglitazone and metformin twice a day (before breakfast and before dinner) orally for 12 weeks.
  Interventions: Drug: Pioglitazone and Metformin
- Placebo (Placebo Comparator): Type 2 diabetic patients only took SUs previously. During a week for washout before the trial, they received diet and sport instructions, kept the SUs unchanged and didn't use any drugs affecting blood glucose. All participants added 1 tablet of placebo twice a day (before breakfast and before dinner) orally for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone and Metformin — taking 1 tablet twice a day (before breakfast and before dinner) orally for 12 weeks
  Other Names: Compound Preparation of Pioglitazone and Metformin; Kashuangping; H20100180
  Arms: Pioglitazone and Metformin
Drug: Placebo — taking 1 tablet twice a day (before breakfast and before dinner) orally for 12 weeks
  Arms: Placebo

SUMMARY:
Secondary failure of sulfonylureas (SUs) can occur in about 30%-40% of type 2 diabetic patients after treatment with SUs for 5 years, although SUs are widely used in type 2 diabetic patients. This study was designed to evaluate the effectiveness and safety of adding compound preparation of pioglitazone and metformin for type 2 diabetic patients who have bad glycemic control with the initial treatment of SUs.

DETAILED DESCRIPTION:
Design of this clinical trial was multicenter, randomized, double-blind and placebo parallel controlled. Type 2 diabetic patients having bad glycemic control with the initial treatment of SUs were included. They were randomly divided into experiment group and control group, respectively taking compound preparation of pioglitazone and metformin (2mg/500mg) and placebo with identical shape immediately before a meal twice a day. Course of the treatment was 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients (WHO criterion, 1999)
* 19kg/m2 ≤ BMI ≤ 35kg/m2
* Subject with the initial treatment of SUs on the basis of controlling diet and sport; treatment lasting for no less than 3 months and stable dose for at least 1 month; HbA1c 7-11%
* No insulin therapy during 6 months before being selected
* Not involved in any drug test during 3 months before being selected
* No serious heart, liver or kidney diseases
* Must have effective contraception methods for women of child-bearing age
* Willing to being informed consent

Exclusion Criteria:

* Type 1 diabetes or other specific types of diabetes
* Pregnancy, preparation for pregnancy, lactation and women of child-bearing age incapable of effective contraception methods
* Uncooperative subject because of various reasons
* Abnormal liver function, glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST) > twice the upper limits of normal
* Impairment of renal function, serum creatinine: ≥ 133mmol/L for female，≥ 135mmol/L for male
* Serious chronic gastrointestinal diseases
* Edema
* Serious heart diseases, such as cardiac insufficiency (level III or more according to NYHA), acute coronary syndrome and old myocardial infraction
* Blood pressure: Systolic blood pressure (SBP) ≥ 180mmHg and/or diastolic blood pressure (DBP) ≥ 110mmHg
* White blood count (WBC) < 4.0×109/L or platelet count (PLT) < 90×109/L，or definite anemia (Hb：< 120g/L for male, < 110g/L for female), or other hematological diseases
* Endocrine system diseases, such as hyperthyroidism and hypercortisolism
* Experimental drug allergy or frequent hypoglycemia
* Psychiatric disorders, drug or other substance abuse
* Diabetic ketoacidosis and hyperosmolar nonketotic coma requiring insulin therapy
* Stressful situations such as surgery, serious trauma and so on
* Chronic hypoxic diseases such as pulmonary emphysema and pulmonary heart disease
* Combined use of drugs effecting glucose metabolism such as glucocorticoid
* Tumor, especially bladder tumor and/or family history of bladder tumor and/or long-term hematuria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng Yu, MD, PhD, Principal Investigator — Division of Endocrinology, Tongji Hospital, Huazhong University of Science & Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 participants were recruited at 15 hospitals in Wuhan between March 2012 and September 2013.
Pre-assignment Details: All participants were randomized to the two groups.They had a week for washout before the trial, during which they received diet and sport instructions, kept the sulfonylureas (SUs) unchanged and didn't use any drugs affecting blood glucose.
Period: Overall Study
Arm/Group | Pioglitazone and Metformin | Placebo
Started | 47 | 51
Completed | 43 | 49
Not Completed | 4 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Based on the full analysis set: all participants who were eligible or drop-out, but eliminated participants were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone and Metformin | Placebo | Total
Number analyzed (Participants) | 46 | 51 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.65 (9.91) | 54.51 (7.23) | 54.61 (8.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 26 | 39
  Male | 33 | 25 | 58
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 45 | 50 | 95
  Other ethnicity | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  China | 46 | 51 | 97
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] | 4.86 (3.67) | 4.39 (3.63) | 4.64 (3.63)
Systolic Blood Pressure(SBP) [Mean (Standard Deviation); unit: mmHg] | 125.35 (9.46) | 128.46 (10.38) | 126.86 (9.98)
Diastolic Blood Pressure(DBP) [Mean (Standard Deviation); unit: mmHg] | 76.24 (6.38) | 77.83 (8.78) | 76.87 (7.86)
Height(Male) [Mean (Standard Deviation); unit: cm] | 169.17 (5.03) | 169.92 (6.44) | 169.49 (5.69)
Height(Female) [Mean (Standard Deviation); unit: cm] | 158.23 (6.00) | 159.88 (5.54) | 159.33 (5.68)
Weight(Male) [Mean (Standard Deviation); unit: Kg] | 71.18 (8.03) | 73.37 (10.89) | 72.05 (9.39)
Weight(Female) [Mean (Standard Deviation); unit: Kg] | 64.85 (5.49) | 63.00 (5.49) | 63.62 (5.49)
ln(Fasting Plasma Glucose(FPG)) [Mean (Standard Deviation); unit: ln(mmol/L)] | 2.16 (0.23) | 2.08 (0.18) | 2.12 (0.21)
2-hour Postprandial Glucose(2hPPG) [Mean (Standard Deviation); unit: mmol/L] | 16.47 (3.96) | 15.59 (3.81) | 16.02 (3.86)
ln(HbA1c) [Mean (Standard Deviation); unit: ln(percent)] | 2.14 (0.12) | 2.10 (0.14) | 2.12 (0.19)
ln(Fasting Insulin) [Mean (Standard Deviation); unit: ln(mU/L)] | 2.21 (0.62) | 2.17 (0.58) | 2.19 (0.60)
ln(2-hour Postprandial Insulin) [Mean (Standard Deviation); unit: ln(mU/L)] | 3.49 (0.67) | 3.48 (0.65) | 3.49 (0.66)
Total Cholesterol(TC) [Mean (Standard Deviation); unit: mmol/L] | 4.76 (0.79) | 4.76 (1.04) | 4.76 (0.92)
Triglyceride(TG) [Mean (Standard Deviation); unit: mmol/L] | 1.76 (0.93) | 1.71 (0.90) | 1.74 (0.91)
High Density Lipoprotein(HDL) [Mean (Standard Deviation); unit: mmol/L] | 1.22 (0.25) | 1.13 (0.22) | 1.17 (0.24)
ln(Low Density Lipoprotein(LDL)) [Mean (Standard Deviation); unit: ln(mmol/L)] | 0.90 (0.32) | 0.87 (0.45) | 0.88 (0.39)
Glutamic-pyruvic Transaminase(ALT) [Mean (Standard Deviation); unit: U/L] | 21.98 (8.57) | 25.35 (12.00) | 23.75 (10.60)
Glutamic-oxaloacetic Transaminase(AST) [Mean (Standard Deviation); unit: U/L] | 20.47 (6.92) | 22.25 (7.82) | 21.42 (7.43)
Total Bilirubin(TBil) [Mean (Standard Deviation); unit: mmol/L] | 15.26 (5.87) | 14.09 (5.00) | 14.64 (5.42)
Direct Bilirubin(DBil) [Mean (Standard Deviation); unit: mmol/L] | 3.91 (1.79) | 3.92 (2.11) | 3.92 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Change of HbA1c From Baseline at Week 12
Description: Measuring venous level of HbA1c at the start of the trail and at week 12 in all subjects, then using the natural logarithm of HbA1c to analyze the change in HbA1c from baseline at week 12 and compare that between experiment group and control group, since the HbA1c wasn't normal distribution and was logarithmic normal distribution. Change = ln(Baseline Level) - ln(Week 12 Level).
Time Frame: Baseline, Week 12
Population: Based on the full analysis set: all participants who were eligible or drop-out, but eliminated participants were excluded. Intention to treat analysis and last observational carried forward(LOCF) imputation method.
Measure: Mean (Standard Deviation); unit: ln(percent)
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
ln(percent)
  ln(HbA1c) at Baseline | 2.14 (0.12) | 2.10 (0.14)
  ln(HbA1c) at Week 12 | 1.95 (0.12) | 2.02 (0.17)
  Change from Baseline at Week 12 | 0.19 (0.14) | 0.07 (0.21)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of HbA1c between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance is 0.05; the change was statistical significant with P-value less than 0.05
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of HbA1c between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0650, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of HbA1c between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change of FPG From Baseline at Week 12
Description: Measuring venous level of FPG(fasting plasma glucose) at the start of the trail and at week 12 in all subjects, then using the natural logarithm of FPG to analyze the change in FPG from baseline at week 12 and compare that between experiment group and control group, since the FPG wasn't normal distribution and was logarithmic normal distribution. Change = ln(Baseline Level) - ln(Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ln(mmol/L)
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
ln(mmol/L)
  ln(FPG) at Baseline | 2.16 (0.23) | 2.08 (0.18)
  ln(FPG) at Week 12 | 1.91 (0.22) | 2.05 (0.29)
  Change from Baseline at Week 12 | 0.25 (0.24) | 0.04 (0.28)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of FPG between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of FPG between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0849, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of FPG between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0005, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change of 2hPPG From Baseline at Week 12
Description: Measuring venous level of 2hPPG(2-hour postprandial glucose) at the start of the trail and at week 12 in all subjects, then analyzing the change in 2hPPG from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  2hPPG at Baseline | 16.47 (3.96) | 15.59 (3.81)
  2hPPG at Week 12 | 12.68 (3.43) | 15.23 (3.80)
  Change from Baseline at Week 12 | 3.65 (3.73) | 0.45 (3.94)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of 2hPPG between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of 2hPPG between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.2428, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of 2hPPG between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0003, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change of Fasting Insulin From Baseline at Week 12
Description: Measuring venous level of fasting insulin at the start of the trail and at week 12 in all subjects, then using the natural logarithm of fasting insulin to analyze the change in fasting insulin from baseline at week 12 and compare that between experiment group and control group, since the fasting insulin wasn't normal distribution and was logarithmic normal distribution. Change = ln(Baseline Level) - ln(Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ln(mU/L)
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
ln(mU/L)
  ln(Fasting Insulin) at Baseline | 2.21 (0.62) | 2.17 (0.58)
  ln(Fasting Insulin) at Week 12 | 1.90 (0.58) | 2.26 (0.74)
  Change from Baseline at Week 12 | 0.35 (0.58) | -0.08 (0.79)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of fasting insulin between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of fasting insulin between before and after treatment in Placebo group.. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.7353, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of fasting insulin between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0013, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change of 2-hour Postprandial Insulin From Baseline at Week 12
Description: Measuring venous level of 2-hour postprandial insulin at the start of the trail and at week 12 in all subjects, then using the natural logarithm of 2-hour postprandial insulin to analyze the change in 2-hour postprandial insulin from baseline at week 12 and compare that between experiment group and control group, since the 2-hour postprandial insulin wasn't normal distribution and was logarithmic normal distribution. Change = ln(Baseline Level) - ln(Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ln(mU/L)
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
ln(mU/L)
  ln(2-hour Postprandial Insulin) at Baseline | 3.49 (0.67) | 3.48 (0.65)
  ln(2-hour Postprandial Insulin) at Week 12 | 3.33 (0.75) | 3.64 (0.74)
  Change from Baseline at Week 12 | 0.19 (0.83) | -0.15 (0.77)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of 2-hour postprandial insulin between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.1147, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of 2-hour postprandial insulin between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.4006, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of 2-hour postprandial insulin between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0614, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change of TC From Baseline at Week 12
Description: Measuring venous level of TC(Total Cholesterol) at the start of the trail and at week 12 in all subjects, then analyzing the change in TC from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  TC at Baseline | 4.76 (0.79) | 4.76 (1.04)
  TC at Week 12 | 4.74 (0.88) | 4.66 (0.83)
  Change from Baseline at Week 12 | 0.06 (0.60) | 0.09 (0.80)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of TC between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3795, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of TC between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.4236, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of TC between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change of TG From Baseline at Week 12
Description: Measuring venous level of TG(Triglyceride) at the start of the trail and at week 12 in all subjects, then analyzing the change in TG from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  TG at Baseline | 1.76 (0.93) | 1.71 (0.90)
  TG at Week 12 | 1.66 (0.94) | 1.85 (1.49)
  Change from Baseline at Week 12 | 0.09 (0.77) | -0.17 (1.24)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of TG between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3151, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of TG between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.6963, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of TG between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3204, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change of HDL From Baseline at Week 12
Description: Measuring venous level of HDL(High-Density Lipoprotein) at the start of the trail and at week 12 in all subjects, then analyzing the change in HDL from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  HDL at Baseline | 1.22 (0.25) | 1.13 (0.22)
  HDL at Week 12 | 1.33 (0.29) | 1.15 (0.26)
  Change from Baseline at Week 12 | -0.09 (0.19) | 0.00 (0.17)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of HDL between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0038, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of HDL between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3812, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of HDL between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0108, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change of LDL From Baseline at Week 12
Description: Measuring venous level of LDL(Low-Density Lipoprotein) at the start of the trail and at week 12 in all subjects, then using the natural logarithm of LDL to analyze the change in LDL from baseline at week 12 and compare that between experiment group and control group, since the LDL wasn't normal distribution and was logarithmic normal distribution. Change = ln(Baseline Level) - ln(Week 12 Level).
Time Frame: Baseline, Week 12
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: ln(mmol/L)
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
ln(mmol/L)
  ln(LDL) at Baseline | 0.90 (0.32) | 0.87 (0.45)
  ln(LDL) at Week 12 | 0.89 (0.28) | 0.83 (0.34)
  Change from Baseline at Week 12 | 0.02 (0.20) | 0.03 (0.42)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of LDL between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.5476, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of LDL between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.1248, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of LDL between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3620, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

10. Other Pre Specified Outcome: Change of ALT From Baseline at Week 12
Description: Measuring venous level of ALT at the start of the trail and at week 12 in all subjects, then analyzing the change in ALT from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: Based on safety set：all participants who received intervention at least once and had actual data of safety record.
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
U/L
  ALT at Baseline | 21.98 (8.57) | 25.35 (12.00)
  ALT at Week 12 | 21.63 (7.17) | 24.80 (10.01)
  Change from Baseline at Week 12 | 0.40 (9.14) | 0.47 (13.88)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of ALT between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.5636, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of ALT between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.3681, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of ALT between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.2589, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

11. Other Pre Specified Outcome: Change of AST From Baseline at Week 12
Description: Measuring venous level of AST at the start of the trail and at week 12 in all subjects, then analyzing the change in AST from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: Based on safety set：all participants who received intervention at least once and had actual data of safety record.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
U/L
  AST at Baseline | 20.47 (6.92) | 22.25 (7.82)
  AST at Week 12 | 21.12 (5.58) | 21.87 (6.03)
  Change from Baseline at Week 12 | -0.41 (7.35) | 0.41 (8.50)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of AST between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.7972, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of AST between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.7801, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of AST between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.8744, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

12. Other Pre Specified Outcome: Change of TBil From Baseline at Week 12
Description: Measuring venous level of TBil(total bilirubin) at the start of the trail and at week 12 in all subjects, then analyzing the change in TBil from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: Based on safety set：all participants who received intervention at least once and had actual data of safety record.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  TBil at Baseline | 15.26 (5.87) | 14.09 (5.00)
  TBil at Week 12 | 14.72 (6.09) | 13.44 (4.23)
  Change from Baseline at Week 12 | 0.31 (6.53) | 0.57 (4.65)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; Null hypothesis is that there was no difference in change of DBil between before and after treatment in Pioglitazone and Metformin group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.8034, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of TBil between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.7675, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of TBil between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.6918, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

13. Other Pre Specified Outcome: Change of DBil From Baseline at Week 12
Description: Measuring venous level of DBil(direct bilirubin) at the start of the trail and at week 12 in all subjects, then analyzing the change in DBil from baseline at week 12 and comparing that between experiment group and control group. Change = (Baseline Level - Week 12 Level).
Time Frame: Baseline, Week 12
Population: Based on safety set：all participants who received intervention at least once and had actual data of safety record.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone and Metformin | Placebo
Number analyzed (Participants) | 46 | 51
mmol/L
  DBil at Baseline | 3.91 (1.79) | 3.92 (2.11)
  DBil at Week 12 | 3.69 (2.08) | 3.32 (1.15)
  Change from Baseline at Week 12 | 0.12 (2.08) | 0.55 (2.04)
Statistical Analysis 1: Comparison: Pioglitazone and Metformin; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0339, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo; Null hypothesis is that there was no difference in change of DBil between before and after treatment in Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.0997, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pioglitazone and Metformin vs Placebo; Null hypothesis is that there was no difference in change of DBil between Pioglitazone and Metformin group and Placebo group. The test was performed with a significance level of 0.05; Test type: Superiority or Other; p = 0.5015, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Safety set included all participants who received intervention at least once and had the actual data of safety index.
Arm/Group | Pioglitazone and Metformin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/51
Other Adverse Events (participants affected / at risk) | 7/46 | 5/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone and Metformin (N=47) | Placebo (N=51)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) — The only death caused by sudden stroke had no clinical association with the drug and wasn't included in safety set. So the total number of participants at risk for serious adverse events in experiment group was 47 rather than 46.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone and Metformin (N=46) | Placebo (N=51)
Hypoglycemia (Endocrine disorders) | 1 (1) | 2 (2) — The total number of participants at risk for other adverse events in experiment group was 46 based on safety set.
Abnormal Liver Function (Hepatobiliary disorders) | 6 (6) | 3 (3) — 6 participants in experiment group and 3 participants in control group had mildly abnormal liver functions at week 12, but these abnormities had no clinical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes